CLINICAL TRIAL: NCT01912222
Title: A Phase 1 Pharmacokinetic Study of Oral IXAZOMIB (MLN9708) in Patients With Advanced Solid Tumors or Hematologic Malignancies With Varying Degrees of Liver Dysfunction
Brief Title: Pharmacokinetic Study of Oral IXAZOMIB in Cancer Patients With Liver Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C16018; U1111-1177-7929 (Registry Identifier: WHO)
Record Dates: First submitted 2013-07-26; First posted 2013-07-31 (Estimated); Results first posted 2016-03-25 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-02

CONDITIONS: Advanced Solid Tumors; Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IXAZOMIB Arm 1 (Experimental): Experimental: Arm 1 (Normal hepatic function) In the 15 day period that constitutes Part A of the trial, patients will receive a single oral 4 mg dose of IXAZOMIB capsule on Day 1.
  Patients from Part A will then have the option of continuing the study by participating in Part B, starting immediately after Part A, where they will receive IXAZOMIB on Days 1, 8, and 15 of a 28-day cycle
  Interventions: Drug: IXAZOMIB
- IXAZOMIB Arm 2 (Experimental): Experimental: Arm 2 (Moderate hepatic impairment) In the 15 day period that constitutes Part A of the trial, patients will receive a single oral 2.3 mg dose of IXAZOMIB capsule on Day 1.
  Patients from Part A will then have the option of continuing the study by participating in Part B, starting immediately after Part A, where they will receive IXAZOMIB on Days 1, 8, and 15 of a 28-day cycle
  Interventions: Drug: IXAZOMIB
- IXAZOMIB Arm 3 (Experimental): Experimental: Arm 3 (Severe hepatic impairment) In the 15 day period that constitutes Part A of the trial, patients will receive a single oral 1.5 mg dose of IXAZOMIB capsule on Day 1.
  Patients from Part A will then have the option of continuing the study by participating in Part B, starting immediately after Part A, where they will receive IXAZOMIB on Days 1, 8, and 15 of a 28-day cycle
  Interventions: Drug: IXAZOMIB

INTERVENTIONS:
Drug: IXAZOMIB

SUMMARY:
This is a phase 1, 2-part, pharmacokinetic study in patients with advanced solid tumors or hematologic malignancies and varying degrees of liver dysfunction (normal function, moderate hepatic impairement or severe hepatic impairment) as defined by the National Cancer Institute (NCI) Organ Dysfunction Working Group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patients must have a diagnosis of an advanced malignant solid tumor or hematologic malignancy for which standard, curative, or life-prolonging treatment does not exist or is no longer effective
* Total bilirubin and aspartate aminotransferase (AST) levels consistent with normal hepatic function (total bilirubin and AST ≤ the upper limit of normal), moderate hepatic impairment (total bilirubin > 1.5 to 3x the upper limit of normal with any AST level) or severe hepatic impairment (total bilirubin > 3x the upper limit of normal with any AST level)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Female patients who are postmenopausal for at least 1 year OR are surgically sterile OR if of childbearing potential, agree to practice 2 effective methods of contraception at the same time during the entire study through 90 days after the last dose of study drug OR agree to practice true abstinence
* Male patients who agree to practice effective barrier contraception during the entire study and through 90 days after the last dose of study drug OR agree to practice true abstinence
* Voluntary written consent
* Suitable venous access for the conduct of blood sampling
* Appropriate clinical laboratory values as specified in the protocol

Exclusion Criteria:

* Systemic treatment with strong and moderate inhibitors of CYP1A2, strong and moderate inhibitors of CYP3A, or clinically significant CYP3A inducers or use of Ginkgo biloba or St. John's wort within 14 days before the first dose of study drug
* Use of any nicotine-containing products within 14 days before the first dose of study drug
* Central Nervous System Involvement or Symptomatic brain metastasis. Patients with brain metastases: must have stable neurologic status following local therapy (surgery or radiation) for at least 2 weeks after completion of the definitive therapy; and must be without neurologic dysfunction that would confound the evaluation of neurologic and other AEs
* Female patients who are lactating or breastfeeding or have a positive serum pregnancy test
* Serious medical or psychiatric illness that could interfere with participation in the study
* Treatment with any investigational products or radiotherapy within 21 days before the first dose of study drug
* Systemic anticancer therapy within 14 days before the first dose of study drug
* Exposure to nitrosoureas or mitomycin C within 6 weeks before the first dose of study drug
* Treatment with therapeutic monoclonal antibodies or antibody-drug conjugates within 60 days before the first dose of study drug
* Radiotherapy or major surgery within the 14 days preceding the first dose of study drug
* Infection requiring systemic intravenous antibiotic therapy or other serious infection within 14 days before the first dose of study drug
* Life-threatening illness unrelated to cancer
* Severe CNS, pulmonary, or renal disease not related to the patient's cancer
* Known human immunodeficiency virus (HIV) positive
* Evidence of uncontrolled cardiovascular conditions
* QTc > 500 milliseconds (msec) on a 12-lead ECG obtained during the Screening period
* Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of IXAZOMIB
* Known allergy to the study medication, its analogues, or excipients in the formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Fairway, Kansas
  - Cleveland, Ohio
  - Dallas, Texas
  - Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in the United States from 27 August 2013 to 25 March 2015.
Pre-assignment Details: Participants with diagnosis of advanced solid tumors or hematologic malignancies having varying degrees of liver dysfunction enrolled in 1 of 3 treatment groups to receive ixazomib 4 mg (normal hepatic function), 2.3 mg (moderate impairment), 1.5 mg (severe impairment) on Day 1 (Part A, 15 day cycle) and on Days 1,8 and 15(Part B, 28 day cycle).
Groups:
- Normal Hepatic Function (Ixazomib 4 mg): Ixazomib 4 mg, capsule, orally, on Day 1 in the pharmacokinetic part (Part A, 15-day cycle) and once on Days 1, 8 and 15 in the 28 day treatment cycle part (Part B) in participants with normal hepatic function.
- Moderate Hepatic Impairment (Ixazomib 2.3 mg): Ixazomib 2.3 mg, capsule, orally, on Day 1 in the pharmacokinetic part (Part A, 15-day cycle) and once on Days 1, 8 and 15 in the 28 day treatment cycle part (Part B) in participants with moderate hepatic impairment.
- Severe Hepatic Impairment (Ixazomib 1.5 mg): Ixazomib 1.5 mg, capsule, orally, on Day 1 in the pharmacokinetic part (Part A, 15-day cycle) and once on Days 1, 8 and 15 in the 28 day treatment cycle part (Part B) in participants with severe hepatic impairment.
Period: Part A: Pharmacokinetic Period
Arm/Group | Normal Hepatic Function (Ixazomib 4 mg) | Moderate Hepatic Impairment (Ixazomib 2.3 mg) | Severe Hepatic Impairment (Ixazomib 1.5 mg)
Started | 13 | 15 | 20
Completed | 12 | 13 | 18
Not Completed | 1 | 2 | 2
Not completed — Not evaluable for PK analyses | 1 | 2 | 2
Period: Part B: Treatment Period
Arm/Group | Normal Hepatic Function (Ixazomib 4 mg) | Moderate Hepatic Impairment (Ixazomib 2.3 mg) | Severe Hepatic Impairment (Ixazomib 1.5 mg)
Started | 13 | 15 | 20
Completed | 0 | 0 | 0
Not Completed | 13 | 15 | 20
Not completed — Progressive disease | 10 | 12 | 15
Not completed — Adverse Event | 1 | 2 | 3
Not completed — Withdrawal by Subject | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis population was defined as participants who received at least 1 dose of ixazomib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Hepatic Function (Ixazomib 4 mg) | Moderate Hepatic Impairment (Ixazomib 2.3 mg) | Severe Hepatic Impairment (Ixazomib 1.5 mg) | Total
Number analyzed (Participants) | 13 | 15 | 20 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (15.19) | 56.2 (15.26) | 54.5 (13.84) | 56.2 (14.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 6 | 20
  Male | 6 | 8 | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 0 | 4
  Not Hispanic or Latino | 10 | 9 | 20 | 39
  Unknown or Not Reported | 3 | 2 | 0 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  White | 11 | 8 | 13 | 32
  Black or African American | 2 | 2 | 6 | 10
  Other | 0 | 4 | 0 | 4
  Asian | 0 | 1 | 1 | 2
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 168.6 (6.79) | 168.6 (12.56) | 169.6 (27.54) | 169.0 (19.01)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 74.42 (16.788) | 76.97 (12.050) | 76.94 (23.498) | 76.27 (18.431)
Disease type at diagnosis [Number; unit: participants] — Solid tumor includes colon, colorectal, endometrial, esophageal, gall bladder, head and neck, kidney, liver, melanoma, mesothelioma, non-small cell lung cancer, ovarian, pancreatic, prostate, rectal, and sarcoma. Other tumor includes cholangiocarcinoma, malignant fibrous histiocytoma, metastatic poorly differentiated squamous cell carcinoma of the pelvis, moderately differentiated adenocarcinoma compatible with intrahepatic cholangiocarcinoma, unknown primary with liver metastasis, and peritoneal adenocarcinoma.
  participants
    Solid tumor | 10 | 14 | 18 | 42
    Other | 3 | 1 | 2 | 6
Months from initial diagnosis to first dose of ixazomib [Mean (Standard Deviation); unit: months] | 56.5 (43.40) | 23.7 (16.59) | 35.2 (28.73) | 37.4 (32.56)
Participants with prior antineoplastic therapy [Number; unit: participants] — All participants had prior antineoplastic therapy.
  participants | 13 | 15 | 20 | 48
Participant with prior radiation [Number; unit: participants]
  Had prior radiation | 6 | 6 | 11 | 23
  Had no prior radiation | 7 | 9 | 9 | 25
Participant with prior surgery [Number; unit: participants]
  Had prior surgery | 12 | 14 | 18 | 44
  Had no prior surgery | 1 | 1 | 2 | 4
Baseline Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — ECOG assessed participant's performance status on 5 point scale: 0=Fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory (>50% of waking hrs), capable of all self care, unable to carry out any work activities; 3=capable of only limited self care, confined to bed/chair >50% of waking hrs; 4=completely disabled, cannot carry on any self care, totally confined to bed/chair; 5=dead. Participants who had a score of 0 or 1 were assessed.
  participants
    0 | 1 | 0 | 1 | 2
    1 | 12 | 15 | 19 | 46
Baseline total bilirubin [Mean (Standard Deviation); unit: micro mole per liter (mcmol/L)] | 7.43 (3.092) | 40.25 (5.594) | 108.61 (78.372) | 59.85 (66.249)
Baseline aspartate aminotransferase (AST) [Mean (Standard Deviation); unit: units per liter (U/L)] | 21.04 (6.884) | 169.97 (147.433) | 197.48 (198.211) | 141.09 (167.256)

OUTCOME MEASURES:

1. Primary Outcome: Unbound AUC(0-last): Unbound Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Ixazomib
Time Frame: Part A, Day 1: Pre-dose and at multiple timepoints (up to 336 hours) post-dose
Population: The PK analysis population was defined as participants who received the single dose of ixazomib in Part A of the study, did not receive any excluded concomitant medications through the completion of PK sampling, and had sufficient concentration-time data to permit the reliable estimation of PK parameters by noncompartmental analysis methods.
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hours per milliliter (ng*hr/mL)
Arm/Group | Normal Hepatic Function (Ixazomib 4 mg) | Moderate Hepatic Impairment (Ixazomib 2.3 mg) | Severe Hepatic Impairment (Ixazomib 1.5 mg)
Number analyzed (Participants) | 12 | 10 | 11
nanogram*hours per milliliter (ng*hr/mL) | 9.6476 (5.39885) | 7.3292 (5.35269) | 4.4383 (4.21266)

2. Primary Outcome: Unbound Cmax: Unbound Maximum Observed Plasma Concentration for Ixazomib
Time Frame: Part A, Day 1: Pre-dose and at multiple timepoints (up to 336 hours) post-dose
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Normal Hepatic Function (Ixazomib 4 mg) | Moderate Hepatic Impairment (Ixazomib 2.3 mg) | Severe Hepatic Impairment (Ixazomib 1.5 mg)
Number analyzed (Participants) | 12 | 13 | 18
nanogram per milliliter (ng/mL) | 0.50893 (0.271928) | 0.37245 (0.385113) | 0.23176 (0.271358)

3. Primary Outcome: Tmax- Time to Reach the Maximum Plasma Concentration (Cmax) for Ixazomib
Time Frame: Part A, Day 1: Pre-dose and at multiple timepoints (up to 336 hours) post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Hepatic Function (Ixazomib 4 mg) | Moderate Hepatic Impairment (Ixazomib 2.3 mg) | Severe Hepatic Impairment (Ixazomib 1.5 mg)
Number analyzed (Participants) | 12 | 13 | 18
hours | 0.950 [0.48 to 4.00] | 1.500 [0.50 to 2.50] | 1.205 [0.50 to 4.00]

4. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAE) and Serious Adverse Events (SAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Baseline up to 30 days after last dose of study drug (Day 45 for each treatment cycle for up to a maximum of 12 cycles [28 days treatment cycles])
Population: The safety analysis population was defined as participants who received at least 1 dose of ixazomib.
Measure: Number; unit: participants
Arm/Group | Normal Hepatic Function (Ixazomib 4 mg) | Moderate Hepatic Impairment (Ixazomib 2.3 mg) | Severe Hepatic Impairment (Ixazomib 1.5 mg)
Number analyzed (Participants) | 13 | 15 | 20
participants
  TEAE | 13 | 15 | 20
  SAE | 6 | 10 | 15

5. Primary Outcome: Number of Participants Reporting Clinically Significant Change From Baseline in Laboratory Values
Description: The number of participants with any markedly abnormal standard safety laboratory values collected throughout study.
Time Frame: Baseline up to Day 15 for each treatment cycle (28 days treatment cycle for up to a maximum of 12 cycles)
Population: The safety analysis population was defined as participants who received at least 1 dose of ixazomib.
Measure: Number; unit: participants
Arm/Group | Normal Hepatic Function (Ixazomib 4 mg) | Moderate Hepatic Impairment (Ixazomib 2.3 mg) | Severe Hepatic Impairment (Ixazomib 1.5 mg)
Number analyzed (Participants) | 13 | 15 | 20
participants | 0 | 0 | 0

6. Primary Outcome: Number of Participants Reporting Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs included body temperature (oral or tympanic measurement), sitting blood pressure (after the participant has rested for at least 5 minutes), and pulse (bpm).
Time Frame: Baseline up to Day 15 for each treatment cycle (28 days treatment cycle for up to a maximum of 12 cycles)
Population: The safety analysis population was defined as participants who received at least 1 dose of ixazomib.
Measure: Number; unit: participants
Arm/Group | Normal Hepatic Function (Ixazomib 4 mg) | Moderate Hepatic Impairment (Ixazomib 2.3 mg) | Severe Hepatic Impairment (Ixazomib 1.5 mg)
Number analyzed (Participants) | 13 | 15 | 20
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug (up to cycle 12 [each cycle is 28 days]).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Normal Hepatic Function (Ixazomib 4 mg) | Moderate Hepatic Impairment (Ixazomib 2.3 mg) | Severe Hepatic Impairment (Ixazomib 1.5 mg)
Serious Adverse Events (participants affected / at risk) | 6/13 | 10/15 | 15/20
Other Adverse Events (participants affected / at risk) | 12/13 | 14/15 | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Hepatic Function (Ixazomib 4 mg) (N=13) | Moderate Hepatic Impairment (Ixazomib 2.3 mg) (N=15) | Severe Hepatic Impairment (Ixazomib 1.5 mg) (N=20)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 — The occurrence of this event led to death of one study participant in ixazomib 2.3 mg treatment arm.
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 6 — The occurrence of this event led to death of one study participants in ixazomib 2.3 mg treatment arm and three study participants in ixazomib 1.5 mg treatment arm.
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 1 — The occurrence of this event led to death of one study participant in ixazomib 2.3 mg treatment arm and one study participant in ixazomib 1.5 mg treatment arm.
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 — The occurrence of this event led to death of one study participant in ixazomib 1.5 mg treatment arm.
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Axillary pain (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 — The occurrence of this event led to death of one study participant in ixazomib 1.5 mg treatment arm.
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — The occurrence of this event led to death of one study participant in ixazomib 2.3 mg treatment arm.
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 — The occurrence of this event led to death of one study participant in ixazomib 1.5 mg treatment arm.
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 — The occurrence of this event led to death of one study participant in ixazomib 1.5 mg treatment arm.
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 — The occurrence of this event led to death of one study participant in ixazomib 2.3 mg treatment arm.
Device related infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 — The occurrence of this event led to death of one study participant in ixazomib 2.3 mg treatment arm.
Mental status changes (Psychiatric disorders) | 0 | 0 | 2
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Hepatic Function (Ixazomib 4 mg) (N=13) | Moderate Hepatic Impairment (Ixazomib 2.3 mg) (N=15) | Severe Hepatic Impairment (Ixazomib 1.5 mg) (N=20)
Decreased appetite (Metabolism and nutrition disorders) | 7 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 3
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 2 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 2
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 3
Ammonia increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2
Amylase increased (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 1
Waist circumference increased (Investigations) | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Malaise (General disorders) | 2 | 0 | 1
Chills (General disorders) | 0 | 0 | 1
Early satiety (General disorders) | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Photopsia (Eye disorders) | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.